CLINICAL TRIAL: NCT05196503
Title: Efficacy of Platelet Rich Fibrin in the Prevention of Residual Neuropathic Pain Following Disc Herniation Surgery
Brief Title: Efficacy of an Intraoperative Periradicular Application of Platelet Rich Fibrin (PRF) on the Intensity of Residual Post-surgical Neuropathic Pain After a Surgery for Disc Herniation
Acronym: NeuroPRF
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8363
Record Dates: First submitted 2021-08-26; First posted 2022-01-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Neuropathic Pain; Chronic Postsurgical Pain
Keywords: Neuropathic pain; Chronic postsurgical pain prevention; Intraoperative platelet rich fibrin; Disc herniation surgery
MeSH Terms: conditions — Neuralgia; Pain, Postoperative | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Surgery for disc herniation and intraoperative periradicular administration of PRF
  Interventions: Biological: Treatment
- Control group (Active Comparator): Surgery for disc herniation alone (i.e. reference treatment).
  Interventions: Biological: Treatment

INTERVENTIONS:
Biological: Treatment — Experimental product: product derived from autologous blood, obtained after centrifugation.
  Treatment modalities: intraoperative periradicular administration of autologous PRF.

SUMMARY:
The prevalence of post-surgical lumbar neuropathic radiculopathy is approximately 30%. Poor response to the treatments recommended for neuropathic pain, namely antidepressants and/or gabapentinoids, requires the development of new techniques to prevent this chronic pain. Certain well-tolerated techniques, such as the administration of plasma enriched with platelets and fibrin (PRF), are increasingly used in regenerative medicine for their anti-inflammatory and analgesic properties. Thus, a periradicular intraoperative application of PRF may have an analgesic effect on the intensity of residual postsurgical neuropathic pain after disc herniation surgery.

DETAILED DESCRIPTION:
A superiority study, phase III, prospective, single-center, randomized in parallel groups and conducted in a single-blind manner, with evaluation by a blind outcome assessor. Patients will be randomized to one of two treatment groups: Experimental group (surgery and periradicular administration of PRF) or Control group (reference treatment, surgery alone).

ELIGIBILITY:
Inclusion criteria:

* Patient, male or female, >18 years old at the time of signing informed consent;
* Patient for whom a diagnosis of radiculopathy on lumbar disc herniation has been made, and for whom surgery has been scheduled in the Neurosurgery department;
* Patient affiliated to a social security health insurance scheme;
* Patient able to understand the objectives and risks of research and to give informed, dated and signed consent;
* Patient having been informed of the results of the prior medical examination;
* Women of childbearing age provided that a negative blood pregnancy test is recorded at the inclusion visit and effective contraception used throughout the study.

Exclusion criteria:

* Patient with a history of lumbar spinal surgery (multiple herniated discs, herniated disc other than lumbar);
* Patient with HIV, active cancer, HBV, HCV (verified by interview);
* Patient on long-term systemic corticosteroid therapy;
* Patient with an ASA score > 3 during the consultation with the anesthesiologist;
* Inability to give the patient informed information (patient in an emergency or life-threatening situation, difficulties in understanding);
* Patient in exclusion period (determined by a previous or ongoing study);
* Subject under safeguard of justice;
* Subject under curatorship;
* Pregnancy;
* Breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Assess the effectiveness of periricular intraoperative application of Platelet- and Fibrin-enriched plasma (PRF) on the intensity of residual neuropathic pain postoperatively with primary herniated disc surgery. | 6 months
  Average intensity, over 24 hours, of a sequellar radicular neuropathic painy an EVA and affirmed by a DN4 score greater than or equal to 4

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires, Strasbourg, Bas-Rhin, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Todeschi J, Dannhoff G, Coca AH, Timbolschi DI, Proust F, Lefebvre F, Lelievre V, Poisbeau P, Vallat L, Salvat E, Bohren Y. Effect of an intraoperative periradicular application of platelet-rich fibrin (PRF) on residual post-surgical neuropathic pain after disc herniation surgery: study protocol for NeuroPRF, a randomized controlled trial. Trials. 2023 Jun 19;24(1):418. doi: 10.1186/s13063-023-07420-y. PMID 37337269